CLINICAL TRIAL: NCT02872818
Title: The Effect of Metformin and Medroxyprogesterone Acetate on Apoptotic Signaling Pathways in Wistar-Albino Rats With Induced Endometrial Hyperplasia
Brief Title: Apoptotic Signaling Pathways in Rats With Endometrial Hyperplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erdem Sahin, Principal Investigator, Kayseri Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14/128
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Apoptotic Signal Pathways in Endometrial Hyperplasia
Keywords: Apoptotic signal pathway; Survivin; Bcl-2; Bax; c-Myc; Caspase-9; endometrial hyperplasia; endometrium cancer
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Metformin; Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (3):
- Control group (Active Comparator): Medicated with only 4mg/kg 17β estradiol hemihydrate for 20 days to develop endometrial hyperplasia
  Interventions: Drug: 17β estradiol hemihydrate
- Metformin group (Active Comparator): Having been obtained hyperplasia, the investigators continued medication with 50 mg/kg metformin in addition to 17β estradiol hemihydrate for 10 days
  Interventions: Drug: 17β estradiol hemihydrate; Drug: Metformin
- Medroxyprogesterone acetate group (Active Comparator): Having been obtained hyperplasia, the investigators continued medication with 1mg/day medroxyprogesterone acetate in addition to 17β estradiol hemihydrate for 10 days
  Interventions: Drug: 17β estradiol hemihydrate; Drug: medroxyprogesterone acetate

INTERVENTIONS:
Drug: 17β estradiol hemihydrate — 4mg/kg/day for 20 days
Drug: Metformin — 50 mg/kg/day last 10 days
  Arms: Metformin group
Drug: medroxyprogesterone acetate — 1mg/kg/day last 10 days
  Arms: Medroxyprogesterone acetate group

SUMMARY:
The purpose of the study is to determine apoptotic signaling pathways such as Survivin, Bcl-2, Bax, c-Myc and caspase-9 expression levels in rats model with iatrogenic endometrial hyperplasia after metformin and medroxyprogesterone acetate administration.

ELIGIBILITY:
Inclusion criteria:

Forty-eight weeks old female Wistar-Albino rats, weighting between 180 and 260 g

Exclusion criteria.

We have no exclusion criteria because we examine drugs effects in the experimental rats

Ages: 8 Weeks to 10 Weeks | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Survivin Gene Expression Levels in Rat Uterine Tissue | 4 months
Bcl-2 Gene Expression Levels in Rat Uterine Tissue | 4 months
Bax Gene Expression Levels in Rat Uterine Tissue | 4 months
c-Myc Gene Expression Levels in Rat Uterine Tissue | 4 months
Caspase-9 Expression Levels in Rat Uterine Tissue | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Erdem SAHİN, Study Director — Kayseri Training and Research Hospital
Locations (1):
- Kayseri Training and Research Hospital, Kayseri, Turkey (Türkiye)